CLINICAL TRIAL: NCT07312565
Title: The Occurrence of Abdominal Aortic Aneurysms in Patients With Ruptured Intracranial Aneurysms
Brief Title: Occurrence of Abdominal Aortic Aneurysms in Patients With Aneurysmal Subarachnoid Hemorrhage
Status: Not yet recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Jeroen J.W.M. Brouwers MD PhD, Principal Investigator, Leiden University Medical Center
Other Study IDs: NL-009714
Record Dates: First submitted 2025-12-02; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Aneurysm Abdominal; Cerebral Aneurysm Ruptured
Keywords: abdominal aortic aneurysm; aneurysmal subarachnoid hemorrhage; ruptured intracranial aneurysm; prospective single cohort study; ultrasound
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with aSAH from the SPARTA trial: All aSAH patients from a large prospective cohort trial in the Netherlands will be screened for eligibility(12). The Study on Prognosis of Acutely RupTured Aneurysms (SPARTA) is an observational prospective cohort trial conducted in the Netherlands in several clinical centres. The aim of this study is to evaluate the long-term clinical outcome of aSAH patients who underwent neurosurgical- or endovascular treatment for their ruptured IA. The study has a population of around 900 patients. Because of the lethality of aSAH, a large proportion of this study population will be diseased or heavily incapacitated.

SUMMARY:
Rationale: Aneurysms of different types are known to be associated. In literature, concurrence of intracranial- and aortic aneurysms is described. Screening for aortic aneurysms (AA) in patients with intracranial aneurysms (IA) or aneurysmal subarachnoid haemorrhage (aSAH) could be cost-effective and of significant importance to decrease morbidity and mortality. The available literature on the association between the two types of aneurysms is sparse and in general of poor methodological quality. This protocol presents a study to more adequately evaluate the association between IA and AA.

Objective: To investigate the occurrence of abdominal aortic aneurysms (AAA) in patients who experienced aSAH.

Study design: This single cohort prospective study will include patients who experienced aSAH. The study participants will receive an abdominal ultrasound of the aorta to detect an AAA.

Study population: aSAH patients from a prospective cohort trial in the Netherlands.

Main study parameters/endpoints: The primary outcome, which will be investigated in the here above described study population, is the number of AAA detected on abdominal ultrasound.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients will not receive an intervention, but only a diagnostic imaging without radiation. The burden associated with this study are considered minimal and the risks negligible. An abdominal ultrasound is a non-invasive diagnostic method with no risks for the participant. The only possible existing burden to the participant is travel and appointment time with a risk of detecting an abdominal aortic aneurysm or other (occult) intra-abdominal pathologies. When an aneurysm, sub-aneurysm or other intra-abdominal pathology is detected, surveillance or treatment according to standard of care and guidelines will follow.

DETAILED DESCRIPTION:
This study will be a prospective single cohort study.

During the period of the study, all aSAH patients (from another prospective cohort trial) will be screened for inclusion eligibility. Eligible patients will be included as subjects in this study. Study subjects will receive an abdominal ultrasound (US) focused on the aorta. Detecting an AAA on abdominal US will result in the daily standard of care for AAA, including surveillance and possible treatment by medication, intervention or surgery.

Study sites This study will be conducted by the Department of Surgery in the main study location University Medical Center Leiden (LUMC) in collaboration with University Neurosurgical Center Holland (UNCH). Eligibility screening and inclusion will be performed by the LUMC.

To answer the research questions of this study, the US laboratory of the LUMC will perform US on the included patients.

The clinical (neurovascular) centers who included patients in the SPARTA trial are:

* Haaglanden Medical Centre (HMC)
* Amsterdam Universitary Medical Centre (AUMC)
* Erasmus Medical Centre (EMC)
* Radboud University Medical Centre (Radboudumc)
* University Medical Centre Utrecht (UMCU)
* Maastricht University Medical Centre (MUMC).

The data from the aortic-scan centers will be obtained and centralized analysis will be performed by the main study location LUMC.

Number of study subjects The investigators will include 233 subjects as one single cohort. In this study, the collected data and analysis will be compared to the general- and at-risk population.

Study duration During an initial period of 2 months, patients will be included as study subjects. Inclusion stops when the targeted number of study subjects (N=233) is reached. The study duration is expected to be around 1.5 years and the study period will end when all 233 study subjects had an abdominal US, or were excluded from the study during the study period for particular reasons.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a participant must meet all of the following criteria:

* Patient is a study subject of the trial: Study on Prognosis of Acutely RupTured Aneurysms (SPARTA)(12)
* Inclusion at least one year after aSAH
* Written informed consent

By being a study subject of the SPARTA trial, the following criteria are applicable:

* Confirmed diagnosis of SAH on CT-scan or lumbar puncture (in the presence of a negative CT-scan)
* IA related SAH as confirmed with radiological imaging
* Age 18 years or older at presentation
* Written informed consent for the SPARTA-trial

Exclusion Criteria:

A potential participant who meets any of the following criteria will be excluded from participation in this study:

* Patient is not a study subject of the SPARTA trial
* Patient has Loeys-Dietz-, Marfan- or Ehlers-Danlos syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All aSAH patients from a large prospective cohort trial in the Netherlands will be screened for eligibility(12). The Study on Prognosis of Acutely RupTured Aneurysms (SPARTA) is an observational prospective cohort trial conducted in the Netherlands in several clinical centres. The aim of this study is to evaluate the long-term clinical outcome of aSAH patients who underwent neurosurgical- or endovascular treatment for their ruptured IA. The study has a population of around 900 patients. Because of the lethality of aSAH, a large proportion of this study population will be diseased or heavily incapacitated.
Sampling Method: Probability Sample
Enrollment: 233 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of AAA | 1 year
  Main study parameter/endpoint The primary endpoint of this study will be the occurrence rate of AAA in the study population. This occurrence rate will be calculated as the proportion of all performed ultrasounds in the study group (N; %).

SECONDARY OUTCOMES:
Risk factors for AAA in aSAH patients | 1 year
  Secondary study parameters/endpoint As a secondary endpoint, the investigators will evaluate risk factors of having an AAA as an aSAH patient. Presence of these factors (i.e. smoking, aneurysmal disease in medical history, age, gender) will be calculated as the proportion of the total study population (N; %).

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Brouwers, MD, PhD, Principal Investigator — Leiden University Medical Centre

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT07312565/Prot_SAP_000.pdf